CLINICAL TRIAL: NCT06371937
Title: Blood Biomarkers From Ethnically Diverse Cardiovascular Patients
Brief Title: iPSC Biobank of Biomarkers Diversity in Cardiovascular Disease
Acronym: INFERENCE
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Greenstone Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Chandy, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 120687
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Arrythmia; Cardiomyopathies; Heart Failure; Cerebrovascular Accident; Congenital Heart Disease; Cardiometabolic Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac; Cardiomyopathies; Heart Failure; Stroke; Heart Defects, Congenital; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The Investigators propose collecting two blood samples of 10 mL each from healthy donors and patients in two tubes containing the anticoagulants heparin and ethylenediaminetetraacetic acid (EDTA), respectively. Blood collection and immediate processing have a higher impact on the results of research and laboratory studies.
  Collected blood samples will be layered over lymphoprep (Stemcell Technologies) in SepMateTM tubes (Stem cell Technologies). Based on density gradient centrifugation the PBMC is isolated by centrifugation, at 2000 rpm for 10 min, transferred, and washed with RPMI media for 5 mins at 1500 rpm. The collected PBMCs are cryopreserved at -196˚C at the C3RP facility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study controls: Healthy control participants (n=50) aged 80 and older enrolled in the study with no known CVD or history of significant medical problems.
- cardiovascular disease: Participants with cardiovascular disease (n=150)

SUMMARY:
The Investigators will create a clinical database and a Biobank of stem cells derived from the blood of participants with cardiovascular disease. The Investigators will recruit participants from diverse racial and ethnic backgrounds with equal representation from both sexes. The Investigators expect to create stem cells and analyze the blood for protein biomarkers and genetic causes of cardiovascular disease. The stem cell biobank and clinical data will be a powerful tool for studying cardiovascular disease.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of morbidity and mortality. The development of cardiovascular disease includes both genetic and epigenetic factors. Understanding their molecular and cellular mechanism is necessary to identify novel drug targets and treat the disease. Present in vitro and in vivo models of the disease do not mimic human pathophysiology, and obtaining the primary cells from the patients for the studies relevant to the cardiovascular and pulmonary system is difficult. Induced pluripotent stem cells (iPSCs) are derived from a person's blood cells and facilitate the discovery of cardiovascular disease mechanisms. The Investigators propose recruiting cardiovascular patients from diverse ethnic backgrounds and creating a rich clinical database using REDCap. Blood samples will be obtained from participants and used to create iPSCs. The participant will have DNA sequencing, and serum will be analyzed for protein biomarkers. The multi-omics data and reprogrammed iPSCs will be stored in the Cardiology and Critical Care (C3RP) laboratory at the Robarts Research Institute at Western University. The reprogrammed iPSCs can generate a limitless supply of cardiovascular tissue. Moreover, the iPSC-derived data will be correlated with clinical information, genetic sequencing, and protein biomarkers from serum analysis. The Investigators expect to create an iPSC biobank coupled with a rich clinical dataset, including genetic sequencing analysis and protein biomarkers that will enable the discovery of novel biomarkers and drug targets for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 to 80 years of age)
* Cardiovascular Disease (CVD)
* Cerebrovascular Disease (CBD)
* Peripheral Vascular Disease (PVD)
* Inherited Arrhythmias
* Cardiomyopathies
* Congenital Heart Disease (CHD)
* Aortopathy
* Hypertension
* Cardiometabolic Disease (CMD)

Exclusion Criteria:

* Younger than 18 years of age.
* Patients not able to provide consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 200 participants including 150 patients with cardiovascular disease and 50 healthy control participants.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2033-06-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
REDCap Database | 10 years
  Identify patients with cardiovascular disease from ethnically diverse backgrounds and create a clinical database with REDCap.
Induced pluripotent stem cell (iPSC) Biobank | 10 years
  Reprogram peripheral blood mononuclear cells (PBMC) to iPSCs.
Differentiation into Cardiovascular lineages | 10 years
  Differentiate of iPSCs into different cardiovascular lineages (endothelial cells, smooth muscle cells, cardiomyocytes, etc.)
Molecular profiling of participants | 10 years
  Molecular profiling of iPSC-derived tissue and patient serum using microarray, DNA sequencing, and high throughput "omics" technologies (transcriptomic analysis, proteomic analysis, metabolomic studies, and functional assays).
Bioinformatics analysis | 10 years
  Bioinformatics analysis of clinical, iPSC disease modeling, and serum omics analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- London Regional Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided